CLINICAL TRIAL: NCT01588925
Title: Hearing Preservation Using Dexamethasone and Hyaluronic Acid for Cochlear Implantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0297/11
Record Dates: First submitted 2012-04-24; First posted 2012-05-01 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2013-03

CONDITIONS: Hearing Loss
Keywords: Cochlear implantation; Dexamethasone; Acid, Hyaluronic
MeSH Terms: conditions — Hearing Loss; Heartburn | interventions — Cochlear Implantation; Dexamethasone; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Experimental): Cochlear Implantation
  Interventions: Device: Cochlear Implantation
- Dexamethasone (Active Comparator): Cochlear implantation using topical dexamethasone
  Interventions: Device: Cochlear Implantation; Drug: Cochlear Implantation+dexamethasone
- Dexamethasone+Hyaluronic acid (Active Comparator): Cochlear implantation using topical dexamethasone associated with hyaluronic acid
  Interventions: Device: Cochlear Implantation; Drug: Cochlear Implantation+dexamethasone+hyaluronic acid

INTERVENTIONS:
Device: Cochlear Implantation — Cochlear implantation using Hybrid L24 Implant
  Other Names: Hybrid L24 Implant
Drug: Cochlear Implantation+dexamethasone — Cochlear implantation using Hybrid L24 Implant,dexamethasone (4mg/ml) in the round window
  Other Names: Hybrid L24 Implant; Dexamethasone (4mg/ml)
  Arms: Dexamethasone
Drug: Cochlear Implantation+dexamethasone+hyaluronic acid — Cochlear implantation using Hybrid L24 Implant,dexamethasone (4mg/ml) in the round window and hyaluronic acid (10mg/ml) in the electrode array
  Other Names: Hybrid L24 Implant; Dexamethasone (4mg/ml); Hyaluronic acid (10mg/ml)
  Arms: Dexamethasone+Hyaluronic acid

SUMMARY:
The objective of the present study is to investigate the effect dexamethasone and hyaluronic acid have on hearing preservation

DETAILED DESCRIPTION:
Many efforts have been made to prevent residual hearing loss after cochlear implantation, such as the development of soft surgical techniques and pharmacological protection.

In this study we investigate whether the topical application of dexamethasone and hyaluronic acid prevents residual hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Adults (greater than 18 years old) with severe/profound, bilateral sensorineural hearing loss with indication of cochlear implantation.
* Hearing thresholds better than 80 dB in 125 Hz, 90 dB in 250Hz and 100 dB in 500, 1000, 2000, 3000 and 4000 Hz in at least 3 of these frequencies

Exclusion Criteria:

* Malformation or cochlear ossification
* Developmental Disabilities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Hearing thresholds | within the first 6 months after surgery
  Hearing thresholds will be measured by audiometry in the frequencies 125, 250, 500, 1000, 2000 and 4000 Hz in the preoperatory, 1 month, 3 months and 6 months after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo F Ramos, Principal Investigator — University of São Paulo General Hospital; Rubens V Brito Neto, Study Director — University of São Paulo General Hospital
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil